CLINICAL TRIAL: NCT07082283
Title: STAPH-CS Study: Short-Term Atrial Pacing and Hemodynamics After Cardiac Surgery - A Prospective Randomized Evaluation of Variable-Rate Atrial Stimulation After Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Short-Term Atrial Pacing and Hemodynamics After Cardiac Surgery
Acronym: STAPH-CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Joanna Tohme, MD, MSc, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEHDF-2702
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Output
Keywords: Cardiopulmonary bypass; Temporary atrial pacing; Pacing frequency; Hemodynamic profile; Cardiac output

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, comparative, single-center study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacing Group (Placebo Comparator): Patients in this group receive continuous atrial pacing at 90 bpm during the first 24 postoperative hours (outside of evaluation sequences).
  Interventions: Procedure: Pacing Protocol for Pacing Group
- Non-Pacing Group (Active Comparator): Patients in this group remain in their spontaneous sinus rhythm outside of the evaluation sequences.
  Interventions: Procedure: Pacing Protocol for Non-pacing Group

INTERVENTIONS:
Procedure: Pacing Protocol for Pacing Group — At four standardized time points (H0: arrival in the ICU, H6, H12, H24), a transient pacing sequence at 70, 80, and 90 bpm is conducted, with each rate applied for 10 minutes to allow stabilization, followed by recording of the hemodynamic profile and blood pressure, as follows:
  * If the patient has a spontaneous rhythm between 50 and 69 bpm, measurements are taken at the spontaneous rate, then at 70 bpm, 80 bpm, and finally 90 bpm
  * If the patient has a spontaneous rhythm between 70 and 79 bpm, measurements are taken at the spontaneous rate, then at 80 bpm, and finally at 90 bpm
  * If the patient has a spontaneous rhythm between 80 and 89 bpm, measurements are taken at the spontaneous rate, then at 90 bpm
  * If the patient has a spontaneous rhythm ≥ 90 bpm, measurements are taken at the spontaneous rate only
  Arms: Pacing Group
Procedure: Pacing Protocol for Non-pacing Group — At H0, H6, H12, and H24, they will undergo transient pacing at 70, 80, and 90 bpm, following the same measurement protocol (10 minutes per rate), followed by recording of the hemodynamic profile and blood pressure, as follows:
  * If the patient has a rhythm between 50 and 69 bpm, measurements will be taken at the spontaneous rate, then at 70 bpm, 80 bpm, and finally 90 bpm
  * If the patient has a rhythm between 70 and 79 bpm, measurements will be taken at the spontaneous rate, then at 80 bpm, and finally at 90 bpm
  * If the patient has a rhythm between 80 and 89 bpm, measurements will be taken at the spontaneous rate, then at 90 bpm
  * If the patient has a rhythm ≥ 90 bpm, measurements will be taken at the spontaneous rate only
  Outside the pacing periods at different rates, patients in the non-pacing group will remain on their spontaneous sinus rhythm.
  Arms: Non-Pacing Group

SUMMARY:
The goal of this clinical trial is to learn whether temporary atrial pacing improves heart function after cardiac surgery under cardiopulmonary bypass (CPB). It will also help determine the best pacing rate during the first 24 hours after surgery. The main questions it aims to answer are:

* Does atrial pacing improve cardiac output after surgery?
* Is 70, 80, or 90 bpm the most effective pacing rate?
* Does pacing reduce the risk of atrial fibrillation after surgery?

DETAILED DESCRIPTION:
Cardiac surgery under cardiopulmonary bypass (CPB) frequently leads to immediate postoperative rhythm or conduction disturbances, especially atrial fibrillation or atrioventricular block (AV Block), along with hemodynamic instability and transient reduction in cardiac output due to myocardial contractility impairment.

Temporary pacing wires are placed in the operating room and have been used since the 1960s to manage cardiac conduction disorders in these patients, allowing for atrial (AAI) or dual-chamber (DDD) pacing if necessary. Atrial pacing, by restoring synchronized atrial contraction with ventricular filling, helps maintain optimal cardiac output.

Cardiac output is defined as the product of heart rate (HR) and stroke volume (SV). To optimize cardiac output, increasing heart rate is possible, hence the need for atrial pacing.

A pacing rate slightly higher than spontaneous sinus rhythm appears to prevent pauses, limit rhythm instability, and reduce the risk of atrial fibrillation. However, the optimal pacing rate postoperatively has not been clearly defined, and data comparing different rates (70, 80, or 90 bpm) are scarce.

In our center, postoperative atrial pacing is nearly routine and commonly set at 90 bpm, a rate we consider optimal due to its alignment with the Frank-Starling curve. This rate maximizes venous return and stroke volume, thereby optimizing postoperative cardiac output.

Nevertheless, several studies have suggested that routine postoperative temporary pacing wire insertion may not always be necessary and should be reserved for patients identified as high-risk for postoperative rhythm disturbances.

Nowadays, in many international centers, the absence of routine temporary pacing has become the norm. Although 90 bpm is theoretically the optimal rate for atrial pacing, important questions remain: Is postoperative pacing absolutely necessary? If so, could a rate lower than 90 bpm suffice to maintain adequate hemodynamic profile (HDP)?

This study aims at determining whether routine temporary pacing is necessary during the first 24 hours after cardiac surgery under CPB, and what the optimal pacing rate is (AAI or DDD: 70 bpm vs. 80 bpm vs. 90 bpm) in terms of its impact on the HDP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Cardiac surgery under CPB (coronary artery bypass grafting, valve replacement or repair, or combined procedures)
* Placement of epicardial atrioventricular pacing wires during surgery
* Placement of a Swan-Ganz catheter intraoperatively
* Signed informed consent

Exclusion Criteria:

* Emergency surgery
* Patients with an internal pacemaker
* History of permanent atrial fibrillation
* Complete atrioventricular block upon weaning from CPB
* Junctional rhythm upon weaning from CPB
* Sinus rhythm < 50 bpm upon weaning from CPB
* Failure of atrial or dual-chamber pacing (patients paced in ventricular mode VVI)
* Contraindication to Swan-Ganz catheter placement
* Hemodynamic instability defined by significant bleeding or tamponade requiring surgical re-intervention, or the need for escalating doses of vasopressors (Norepinephrine > 1 μg/kg/min, Dobutamine > 10 μg/kg/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of different pacing rates on cardiac index measured by Swan-Ganz catheter in the postoperative period following cardiac surgery under cardiopulmonary bypass at H0, H6, H12, and H24. | 24 hours after the surgery
  To evaluate the impact of different pacing rates (50-69 bpm [Category 1], 70-79 bpm [Category 2], 80-89 bpm [Category 3], ≥ 90 bpm [Category 4]) on cardiac index measured by Swan-Ganz catheter in the postoperative period following cardiac surgery under cardiopulmonary bypass (CPB), at H0, H6, H12, and H24.

SECONDARY OUTCOMES:
To determine whether atrial pacing reduces the incidence of atrial fibrillation in the pacing group compared to the non-pacing group in the postoperative period after cardiac surgery under CPB | 24 hours after the surgery
To evaluate the impact of different pacing rates (50-69, 70-79, 80-89, ≥ 90 bpm) on cardiac index measured by Swan-Ganz catheter in patients with heart failure following cardiac surgery under CPB | 24 hours after the surgery
To assess the impact of different pacing rates (50-69, 70-79, 80-89, ≥ 90 bpm) on mean arterial pressure in the postoperative period after cardiac surgery under CPB | 24 hours after the surgery
To evaluate the impact of different pacing rates (50-69, 70-79, 80-89, ≥ 90 bpm) on systemic vascular resistance measured by Swan-Ganz catheter in the postoperative period after cardiac surgery under CPB | 24 hours after the surgery
To assess the impact of different pacing rates (50-69, 70-79, 80-89, ≥ 90 bpm) on stroke volume measured by Swan-Ganz catheter in the postoperative period after cardiac surgery under CPB | 24 hours after the surgery
To evaluate the impact of different pacing rates (50-69, 70-79, 80-89, ≥ 90 bpm) on left and right ventricular work measured by Swan-Ganz catheter in the postoperative period after cardiac surgery under CPB | 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samia Jebara, Study Chair — Saint Joseph University of Beirut
Locations (1):
- Department of Anesthesia and Critical Care, Hôtel-Dieu de France Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No